CLINICAL TRIAL: NCT01189656
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study on Specific-Population to Evaluate the Safety and Efficacy of Therapeutic Double-plasmid HBV DNA Vaccine in HBeAg-positive Patients With Chronic Hepatitis B
Brief Title: A Clinical Study on Therapeutic Double-plasmid Hepatitis B Virus (HBV) DNA Vaccine in Patients With HBeAg-positive Chronic Hepatitis B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The 458 Hospital of Chinese PLA (Other)
Collaborators: Guangzhou Baidi Biotechnology Co., Ltd (Unknown); Guangzhou Pharmaceucal Company Limited (Unknown)
Responsible Party: Guangming Chen, The 458 Hospital of Chinese PLA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71007.02
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Hepatitis B Patients With HBeAg-positive
Keywords: Chronic hepatitis B patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine+Lamivudine group (Experimental): Subjects assigned into the experimental and the controlled groups with randomization and double-blindness by a ratio of 2:1
  Interventions: Biological: HBV DNA Vaccine
- Placebo+Lamivudine group (Placebo Comparator)
  Interventions: Biological: HBV DNA Vaccine

INTERVENTIONS:
Biological: HBV DNA Vaccine — HBV DNA Vaccine, 1mg/ml/syringe, formulation
  Other Names: Therapeutic Double-plasmid HBV DNA Vaccine

SUMMARY:
To preliminarily evaluate the efficiency and safety of therapeutic double- plasmid HBV DNA vaccine on HBeAg-positive, chronic hepatitis B patients, and provide evidence for the next dosing regimen.

DETAILED DESCRIPTION:
The current study is a multicenter, randomized, double-blind, placebo- controlled clinical trial. The eligible subjects are assigned randomly into 2 arms, the Vaccine + Lamivudine group and the Placebo + Lamivudine group, respectively, by a ratio of 2:1. The efficacy variables include the change of HBV DNA load at Week 72, and at each visits the rate of subjects with HBV DNA titer reducing > 2 logarithms ,the change of HBeAg and HBsAg titer, the change of ALT, HBsAg/HBeAg serum conversion rate, the INF-gamma expression level in peripheral blood mononuclear cells (PBMC), the amount of HBV-specific CTL, the change of expression level of peripheral cytokines (IL-4,IL-10,IL-12 and INF-gamma) against the baseline level.

ELIGIBILITY:
Inclusion Criteria:

The following conditions must be met for all enrolled subjects:

1. Aged 18-65 years with either sex;
2. HBV serology meet the following criteria:

   * HBsAg-positive lasting for at least 6 months at the time of screening;
   * HBeAg-positive at the time of screening;
   * Serum HBV DNA≥1.0×10E5 copies/ml at the time of screening
3. 80U/L<ALT<400U/L;
4. TBIL<40μmol/L;
5. No YMDD mutation of the HBV drug resistance gene
6. Subjects agree not to participate in any other clinical trial or take any other anti-HBV therapeutics during the study;
7. Subjects understand and sign the ICF which approved by EC, and are able to comply with the study procedures and complete the study.

Exclusion Criteria:

Subjects meeting the following conditions will not be enrolled in the study:

1. Was suspected with HCC by the following evidence:

   * B-Ultrasound or imaging which shows occupying lesions;
   * Continuingly elevating serum AFP level even if the B-Ultrasound is normal;
   * AFP >100ng/ml;
2. With acute hepatic decompensation caused by liver disease aggravation or with clinical symptoms of decompensated liver disease at baseline;
3. Serum Cr≥1.5mg/dl (≥130μmol/l) at the time of screening;
4. Serum amylase > two-fold of the upper limit of the normal reference value;
5. Hb (male<100g/ L, female<90g/L), WBC<3.5×10E9/L,PLT<60×10E9/L (except hypersplenism and cirrhosis);
6. Co-infection with HCV (anti-HCV positive), HIV and anti-HAV IgM positive, anti-HDV IgM positive, anti-HEV IgM positive, anti-CMV IgM positive and autoimmune hepatitis (e.g. antinuclear antibody titer>1:160 ) or other active liver disease caused by known or unknown factors;
7. Any other serious disease or active diseases other than hepatitis B that are considered by investigators to be potential factors that may interfere with the therapy, assessment or compliance with the protocol, including any uncontrolled diseases with clinical significance, e.g. kidney, heart, lung, blood vessel, neurogenic, digestive system and metabolic diseases (diabetes, hyperthyroidism, adrenal gland diseases), autoimmune dysfunctions, and tumors, etc;
8. History of alcohol or drug abuse that is considered by investigators that could affect subject's compliance with the protocol or could influence the result of the analysis;
9. Pregnant or breast-feeding female subjects, or those who plan to be pregnant during the course of the study or male subjects' companions who plan to be pregnant during the course of the study;
10. Having used immunosuppressive agents, immunomodulators (thymosin), cytotoxic drugs within 6 months or transaminase-decreasing drugs within one month prior to the initiation of this study;
11. Having used anti-HBV drugs (Lamivudine, interferon, adefovir, entecavir, or sebivo, etc.) within 6 months prior to the initiation of this study;
12. Had or planning to have liver transplantation;
13. Having received experimental drug treatment from any other study within 3 months prior to the screening;
14. Allergic to nucleoside drugs or nucleoside analogues;
15. Not agreeing to the study protocol or any other factors considered not eligible for this study by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The change of HBV DNA load at Week 72 | 72 weeks

SECONDARY OUTCOMES:
The rate of subjects with HBV DNA titer reducing > 2 logarithms . | Every 12 weeks
The change of HBeAg and HBsAg titer. | Every 12 weeks
The change of ALT. | Every 12 weeks
HBsAg/HBeAg serum conversion rate. | Every 12 weeks
The INF-gamma expression level in peripheral blood mononuclear cells (PBMC). | Every 12 weeks
The amount of HBV-specific CTL. | Every 12 weeks
The change of expression level of peripheral cytokines (IL-4、IL-10、IL-12 and INF-gamma) against the baseline level. | Every 12 weeks
The different occurence rates of HBV Drug Resistance Gene (YMDD) between the 2 arms. | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yu Yanyan, Professor, Principal Investigator — SFDA
Locations (1):
- Department of Infections Disease of Peking University First Hospital, Beijing, Beijing Municipality, China